CLINICAL TRIAL: NCT01061762
Title: HIV Treatment Adherence Intervention for People With Poor Literacy Skills
Brief Title: Adherence Intervention for People With Low-literacy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Seth Kalichman, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H07-266; R01MH082633-01 (NIH)
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: HIV Infections
Keywords: Treatment adherence; Low literacy skills; HIV treatment
MeSH Terms: conditions — HIV Infections; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Literacy Adherence Counseling (Experimental): 3-counseling sessions for medication adherence improvement tailored for people with poor literacy
  Interventions: Behavioral: Stick To It
- Standard Adherence Counseling (Active Comparator): 3 counseling sessions for adherence improvement derived from standard behavioral approaches.
  Interventions: Behavioral: Standard medication adherence counseling
- Health Counseling Comparison (Active Comparator): 3-sessions of health improvement counseling.
  Interventions: Behavioral: Health Counseling

INTERVENTIONS:
Behavioral: Stick To It — 3-counseling session adherence intervention tailored for people with poor literacy skills
  Arms: Low Literacy Adherence Counseling
Behavioral: Standard medication adherence counseling — 3 counseling sessions for adherence improvement derived from standard behavioral approaches.
  Arms: Standard Adherence Counseling
Behavioral: Health Counseling — 3-session of health improvement counseling to serve as an attention control.
  Arms: Health Counseling Comparison

SUMMARY:
Consistent adherence to antiretroviral therapy is necessary for treatment success. People with poor health literacy skills experience considerable difficulty adhering to their medications. Effective strategies for improving adherence in patients with poor health literacy must be tailored to achieve optimal adherence and therefore viral suppression. This proposal requests support to conduct a randomized clinical trial of a theory-based HIV treatment adherence intervention tailored for people with low-literacy skills.

DETAILED DESCRIPTION:
Adherence to antiretroviral medications is necessary to achieve sufficient HIV suppression and nonadherence can lead to the development of treatment resistant genetic variants of HIV. Research has demonstrated that people living with HIV/AIDS who have low-levels of health literacy experience greater treatment non-adherence than their higher-literacy counterparts. Interventions are urgently needed to improve treatment adherence in people with poor literacy skills. This application proposes to test a theory based behavioral intervention for improving HIV treatment adherence in people living with HIV/AIDS who have low-literacy skills. Grounded in the Information - Motivation - Behavioral Skills (IMB) model of health behavior change, the experimental intervention has been tailored for people with low-levels of health literacy and has been pilot tested in preliminary intervention development research. The intervention is delivered in three one-on-one counseling sessions and one maintenance-focused booster session. The intervention will be conducted in a community care setting in Atlanta. Men and women will be recruited from a AIDS services and infectious disease clinics throughout the Atlanta metropolitan area. Following screening, informed consent and baseline assessments participants will be randomly assigned to receive one of three conditions: (a) Theory-based literacy tailored treatment adherence intervention; (b) standard of care non-tailored time-matched adherence counseling intervention; (c) noncontaminating time-matched attention control intervention. Participants will be followed for 12-months observation. Assessments will include measures of information, motivation, and behavioral skills pertaining to HIV treatment adherence, self-report and objective medication adherence, and viral load. The study will test the hypothesis that a theory-based HIV treatment adherence intervention that is tailored for people with low-literacy will improve HIV treatment adherence and health relative to the standard and attention control conditions. The study will also examine the influence of IMB theoretical constructs on intervention outcomes. The intervention under investigation will be among the first to address treatment adherence among people with poor literacy skills. If shown effective, the intervention model will be ready for immediate dissemination to clinical and community adherence enhancement services for people living with HIV-AIDS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* HIV positive,
* receiving antiretroviral medications, and
* score below cut-off on a standard health literacy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Unannounced Phone Based Pill Counts for Medication Adherence | Baseline, monthly for 12 months

SECONDARY OUTCOMES:
Theoretical Constructs derived from the Information-Motivation-Behavioral Skills Model assessed by psychometric scales of AIDS knowledge, behavioral intentions, adherence self-efficacy, adherence strategies/skills | Baseline, 3, 6, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Seth C Kalichman, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Southeast HIV/AIDS Research and Evaluation Project, Atlanta, Georgia, United States